CLINICAL TRIAL: NCT00724776
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Escalating Single Dose of Albinterferon Alfa 2b (Alb-IFN), Recombinant Human Albumin-interferon Alfa Fusion Protein in Japanese Chronic Hepatitis C Patients.
Brief Title: Albinterferon Alfa 2b Single Dose in Japanese Chronic Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABF656A1202
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2010-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C, Albinterferon alfa 2b, phase I, Japan
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open-label treatment with albinterferon alfa 2b escalating single dose
  Interventions: Biological: Albinterferon alfa 2b

INTERVENTIONS:
Biological: Albinterferon alfa 2b — recombinant human albumin-interferon alfa fusion protein, 600-1800mcg single dose by S.C. on Day 0

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of albinterferon alfa 2b (alb-IFN) single dose in Japanese chronic hepatitis C patients

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of CHC established on the basis of a detectable viral load as measured by a serum HCV RNA test at least 6 months before and during the screening period.
* Age 20 to 69 years
* Have compensated liver disease results on screening laboratory assessment

Exclusion Criteria:

* Evidence of decompensated liver disease and/or liver cirrhosis.
* Body weight < 50 kg.
* A history of immunologically mediated disease.
* A history or other clinical evidence of interstitial lung disease

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after single dose | 5 weeks after single dose

SECONDARY OUTCOMES:
Pharmacokinetics of albinterferon alfa 2b HCV RNA and ALT as pharmacodynamics evaluation | 5 weeks after single dose

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Pharmaceuticals, Japan, Tokyo, Japan

REFERENCES:
- See also: Results for CABF656A1202 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3261